CLINICAL TRIAL: NCT04565119
Title: Biomarkers in the Brain Oxygen Optimization in Severe Traumatic Brain Injury Trial (BioBOOST)
Brief Title: Biomarkers in the Brain Oxygen Optimization in Severe Traumatic Brain Injury Trial
Acronym: BioBOOST
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Michigan (Other); University of Pittsburgh (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 00042151
Record Dates: First submitted 2020-07-01; First posted 2020-09-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: Biomarkers
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum/plasma and CSF samples will be analysed for simultaneous measurement of glial fibrillary acidic protein (GFAP), ubiquitin C-terminal hydrolase L-1 (UCH-L1), tau, and neurofilament light chain (NF-L). These procedures will be carried out in Dr. Diaz-Arrastia's laboratory at the University of Pennsylvania, by a research scientist blinded to the clinical and physiologic data. There will be no difference in the distribution of samples by BOOST-3 treatment group. Other novel brain injury biomarkers will be assayed when they become available. Blood samples collected in the study may be used for both TBI research and the study of other medical conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe traumatic brain injury (TBI): This observational study is ancillary to the Brain Oxygen Optimization in Severe TBI Phase 3 (BOOST-3) trial (NCT 03754114). All participants in Bio-BOOST are enrolled in BOOST-3.
  Interventions: Other: No intervention. This is an observational study.

INTERVENTIONS:
Other: No intervention. This is an observational study. — There are no interventions being tested in the Bio-BOOST study.

SUMMARY:
BioBOOST is a multicenter, observational study of the effect of derangements in brain physiologic parameters on brain injury biomarker levels in patients with severe traumatic brain injury.

DETAILED DESCRIPTION:
This study is a prospective observational, multi-center study of subjects enrolled in the Brain Oxygen Optimization in Severe Traumatic Brain Injury-Phase 3 (BOOST-3) trial. BOOST-3 is a multicenter, randomized, blinded-endpoint, comparative effectiveness study of goal-directed critical care based upon monitoring of brain tissue oxygen and intracranial pressure versus monitoring of intracranial pressure alone in patients with severe traumatic brain injury.

The investigators will obtain an initial set of biospecimens (serum, plasma, cerebrospinal fluid (CSF), DNA and RNA) shortly after randomization into BOOST-3 and within 24 hours of injury. Subsequent biospecimens will be obtained every 8 hours for the first 24 hours post-enrollment. This will allow the characterization of acute changes in biomarker levels. On study days 2 through 5, biospecimens will be obtained twice a day to allow characterization of sub-acute changes in biomarker levels, without overburdening study teams or taking too much blood from individual subjects. On study days 7 and 14 and at 6-months post-enrollment, one set of biospecimen will be obtained, preferably in the morning. Biospecimens collected at each time point will consist of 6 ml of whole blood for serum extraction, 6 ml of whole blood for plasma extraction, 2.5 ml of whole blood for RNA extraction (a total of 14.5 ml [one tablespoon] of blood) and 5 ml of cerebrospinal fluid (CSF).

BioBOOST will utilize data collected in the BOOST-3 trial. This data includes: demographic data and clinical data such as injury characteristics, vital signs, head CT findings, laboratory data and data on physiologic parameters such as intracranial pressure (ICP), partial pressure of brain tissue oxygen (PbtO2), mean arterial pressure (MAP), and cerebral perfusion pressure (CPP), among others.

BioBOOST will also utilize outcome assessment data collected from BOOST-3 participants at 6 months after injury (180 Days ± 30 days). Trained study personnel who are blinded to the treatment arm will administer the outcome assessments, which will include the measures listed below. The battery includes measures of functional status (GOSE), cognition, and emotional health. The 6-month follow-up interview will be done in person whenever possible. It may be done by telephone or video conference with participants where an in-person interview is not possible.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in BOOST-3 (this is an ancillary study to the BOOST-3 trial)
* BOOST-3 participant is enrolled at a BioBOOST site
* Able to maintain initial blood sample within 24 hours of injury
* Provide proxy informed consent

Exclusion Criteria:

* Profoundly anemic (subjects who are profoundly anemic require blood transfusion)
* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to enroll a maximum of 300 male and female subjects among multiple clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak levels of glial fibrillary acidic protein (GFAP) | First 5 days after injury
  This hypothesis will be tested via linear regression model, with peak GFAP level as the response variable and hypoxia exposure as the predictor of interest. Hypoxia exposure will be defined as the depth and duration of PbtO2 < 20 mmHg during the first 48 hours of injury, quantified using area under the curve (AUC) methodology.
Peak levels of ubiquitin C-terminal hydrolase L1 (UCH-L1) | First 5 days after injury
  This hypothesis will be tested via linear regression model, with peak UCH-L1level as the response variable and hypoxia exposure as the predictor of interest. Hypoxia exposure will be defined as the depth and duration of PbtO2 < 20 mmHg during the first 48 hours of injury, quantified using AUC methodology.
Peak levels of neurofilament light chain (NfL) | First 5 days after injury
  This hypothesis will be tested via linear regression model, with peak NfL level as the response variable and hypoxia exposure as the predictor of interest. Hypoxia exposure will be defined as the depth and duration of PbtO2 < 20 mmHg during the first 48 hours of injury, quantified using AUC methodology.
Peak levels of Tau | First 5 days after injury
  This hypothesis will be tested via linear regression model, with peak Tau level as the response variable and hypoxia exposure as the predictor of interest. Hypoxia exposure will be defined as the depth and duration of PbtO2 < 20 mmHg during the first 48 hours of injury, quantified using AUC methodology.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Non-identified IPD will be made available through the Federal Interagency TBI Research (FITBIR) Database.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available upon completion of the study in December of 2026.
Access Criteria: FITBIR qualified investigators will be provided access.

REFERENCES:
- [Background] Okonkwo DO, Shutter LA, Moore C, Temkin NR, Puccio AM, Madden CJ, Andaluz N, Chesnut RM, Bullock MR, Grant GA, McGregor J, Weaver M, Jallo J, LeRoux PD, Moberg D, Barber J, Lazaridis C, Diaz-Arrastia RR. Brain Oxygen Optimization in Severe Traumatic Brain Injury Phase-II: A Phase II Randomized Trial. Crit Care Med. 2017 Nov;45(11):1907-1914. doi: 10.1097/CCM.0000000000002619. PMID 29028696

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT04565119/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT04565119/ICF_001.pdf